CLINICAL TRIAL: NCT01127750
Title: A 4-month, Open-label, Multi-center Study to Explore Tolerability and Safety and Health Outcomes of FTY720 in Patients With Relapsing Forms of Multiple Sclerosis
Brief Title: Tolerability and Safety and Health Outcomes in Relapsing Multiple Sclerosis (MS) Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFTY720D2316; 2010-019029-32 (EudraCT Number)
Record Dates: First submitted 2010-05-19; First posted 2010-05-21 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: Relapsing multiple sclerosis; MS; safety; tolerability; health outcomes
MeSH Terms: interventions — Fingolimod Hydrochloride

ARMS (1):
- FTY720 (Experimental)
  Interventions: Drug: FTY720

INTERVENTIONS:
Drug: FTY720

SUMMARY:
This study will assess tolerability and safety and health outcomes in relapsing MS patients taking FTY720.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age, must have relapsing MS

Exclusion Criteria:

* Patients with a type of MS that is not relapsing
* Patients with history of chronic immune disease
* Patients with a history of certain cancers
* Diabetic patients with certain eye disorders
* Patients who are on certain immunosuppressive medications or heart medications
* Patients with certain heart conditions
* Patients with certain lung conditions

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2417 (Actual)
Dates: Start 2010-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability profile of FTY720 in patients with relapsing forms of MS | 4 months

SECONDARY OUTCOMES:
Incidence of macular edema | 4 months
Incidence of bradyarrhythmic electrocardiograms (ECGs) | 4 months
Patient reported outcomes indices in multiple sclerosis (PRIMUS), short form health survey-12, and treatment satisfaction questionnaire for medication (TSQM-9) | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (230):
- Australia (5):
  - Novartis Investigative Site, Box Hill
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Kogarah
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, Woodville South
- Austria (2):
  - Novartis Investigational Site, Linz
  - Novartis Investigational Site, Vienna
- Belgium (9):
  - Novartis Investigational Site, Bruges
  - Novartis Investigational Site, Brussels
  - Novartis Investigational Site, Charleroi
  - Novartis Investigational Site, Leuven
  - Novartis Investigational Site, Melsbroek
  - Novartis Investigational Site, Overpelt
  - Novartis Investigational Site, Sijsele
  - Novartis Investigational Site, Tinlot
  - Novartis Investigational Site, Wilrijk
- Canada (3):
  - Novartis Investigational Site, Montreal
  - Novartis Investigational Site, Québec
  - Novartis Investigational Site, Victoria
- Czechia (2):
  - Novartis Investigational Site, Prague
  - Novartis Investigational Site, Teplice
- Denmark (2):
  - Novartis Investigational Site, Aarhus
  - Novartis Investigational Site, Copenhagen
- Finland (2):
  - Novartis Investigational Site, Helsinki
  - Novartis Investigational Site, Turku
- Germany (109):
  - Novartis Investigational Site, Aachen
  - Novartis Investigative Site, Aachen
  - Novartis Investigational Site, Aalen
  - Novartis Investigational Site, Abensberg
  - Novartis Investigational Site, Achim
  - Novartis Investigational Site, Alzenau in Unterfranken
  - Novartis Investigational Site, Aschaffenburg
  - Novartis Investigational Site, Attenberg
  - Novartis Investigational Site, Augsburg
  - Novartis Investigational Site, Bad Honnef
  - Novartis Investigational Site, Bad Krozingen
  - Novartis Investigative Site, Bad Mergentheim
  - Novartis Investigational Site, Bad Neustadt / Saale
  - Novartis Investigational Site, Bamberg
  - Novartis Investigative Site, Bayreuth
  - Novartis Investigative Site, Berlin
  - Novarris Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigational Site, Bochum
  - Novartis Investigative Site, Bochum
  - Novaratis Investigative Site, Bochum
  - Novartis Investigational Site, Bogen
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Böblingen
  - Novartis Investigational Site, Braunschweig
  - Novartis Investigational Site, Buchholz
  - Novartis Investigational Site, Chemnitz
  - Novartis Investigative Site, Cologne
  - Novartis Investigational Site, Dillingen
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigational Site, Eisenach
  - Novartis Investigative Site, Emden
  - Novartis Investigational Site, Emmendingen
  - Novartis Investigative Site, Erbach im Odenwald
  - Novartis Investigational Site, Erfurt
  - Novartis Investigational Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigational Site, Essen
  - Novartis Investigational Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigational Site, Greifswald
  - Novartis Investigational Site, Grevenbroich
  - Novartis Investigative Site, Hamburg
  - Novartis Investigational Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigational Site, Herborn
  - Novartis Investigational Site, Herdecke
  - Novartis Investigational Site, Herne
  - Novartis Investigational Site, Homburg
  - Novartis Investigational Site, Itzehoe
  - Novartis Investigational Site, Jena
  - Novartis Investigational Site, Kaltenkirchen
  - Novartis Investigative Site, Kandel
  - Novartis Investigational Site, Karlsruhe
  - Novartis Investigational Site, Karlstadt am Main
  - Novartis Investigational Site, Kassel
  - Neuroscience Research of the Berkshires, Krefeld
  - Novartis Investigational Site, Landshut
  - Novartis Investigational Site, Lappersdorf
  - Novartis Investigational Site, Leipzig
  - Novartis Investigative Site, Lengerich
  - Novartis Investigational Site, Lohr a. Main
  - Novartis Investigational Site, Ludwigshafen
  - Novartis Investigative Site, Ludwigshafen
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mainz
  - Novartis Investigational Site, Mannheim
  - Novartis Investigational Site, Marburg
  - Novartis Investigational Site, Mittweida
  - Novartis Investigational Site, Mönchengladbach
  - Novartis Investigational Site, München
  - Novartis Investigative Site, München
  - Novartis Investigational Site, Münster
  - Novartis Investigational Site, Nagold
  - Novartis Investigational Site, Neu-Ulm
  - Novartis Investigational Site, Neuburg am Inn
  - Novartis Investigational Site, Neuruppin
  - Novartis Investigational Site, Nuremberg
  - Novartis Investigative Site, Oldenburg
  - Novartis Investigational Site, Osnabrück
  - Novartis Investigational Site, Ostfildern
  - Novartis Investigational Site, Pforzheim
  - Novartis Investigational Site, Potsdam
  - Novartis Investigational Site, Prien am Chiemsee
  - Novartis Investigational Site, Regensburg
  - Novartis Investigational Site, Rostock
  - Novartis Investigational Site, Rösrath
  - Novartis Investigative Site, Rüdersdorf
  - Novartis Investigational Site, Schwarzenbruck
  - Novartis Investigative Site, Schwendi
  - Novartis Investigative Site, Siegen
  - Novartis Investigational Site, Sigmaringen
  - Novartis Investigational Site, Sinsheim
  - Novartis Investigative Site, Stade
  - Novartis Investigational Site, Stuttgart
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigational Site, Teupitz
  - Novartis Investigational Site, Tübingen
  - Novartis Investigative Site, Ulm
  - Novartis Investigational Site, Unterhaching
  - Novartis Investigational Site, Wendlingen
  - Novartis Investigational Site, Wermsdorf
  - Novartis Investigational Site, Westerstede
  - Novartis Investigational Site, Wiesbaden
  - Novartis Investigative Site, Wiesbaden
  - Novartis Investigational Site, Wuppertal
  - Novartis Investigational Site, Würzburg
- Greece (3):
  - Novartis Investigational Site, Alexandroupoli
  - Novartis Investigational Site, Athens
  - Novartis Investigational Site, Thessaloniki
- Hungary (3):
  - Novartis Investigational Site, Budapest
  - Novartis Investigational Site, Pécs
  - Novartis Investigational Site, Szeged
- Ireland (2):
  - Novartis Investigational Site, Cork
  - Novartis Investigational Site, Dublin
- Italy (20):
  - Novartis Investigative Site, Acquaviva delle Fonti
  - Novartis Investigative SIte, Asti
  - Novartis Investigative Site, Bergamo
  - Novartis Investigative Site, Bologna
  - Novartis Investigative Site, Cagliari
  - Novartis Investigative Site, Catania
  - Novartis Investigational Site, Foggia
  - Novartis Investigative Site, Foggia
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Napoli
  - Novartis Investigational Site, Napoli
  - Novartis Investigative Site, Palermo
  - Novartis Investigative Site, Pozzilli
  - Novartis Investigative Site, Ravenna
  - Novartis Investigational Site, Roma
  - Novartis Investigative Site, Siena
  - Novartis Investigative Site, Udine
  - Novartis Investigative Site, Verona
  - Novartis Investigative Site, Vicenza
  - Novartis Investigative Site, Viterbo
- Netherlands (6):
  - Novartis Investigational Site, Amsterdam
  - Novartis Investigational Site, Blaricum
  - Novartis Investigational Site, Breda
  - Novartis Investigational Site, Enschede
  - Novartis Investigational Site, Gouda
  - Novartis Investigational Site, Tilburg
- Norway (3):
  - Novartis Investigational Site, Lillehammer
  - Novartis Investigational Site, Molde
  - Novartis Investigational Site, Stavanger
- Poland (3):
  - Novartis Investigational Site, Bydgoszcz
  - Novartis Investigational Site, Katowice
  - Novartis Investigational Site, Lodz
- Portugal (4):
  - Novartis Investigational Site, Amadora
  - Novartis Investigational Site, Coimbra
  - Novartis Investigational Site, Lisbon
  - Novartis Investigational Site, Porto
- Russia (8):
  - Novartis Investigational Site, Kazan'
  - Novartis Investigational Site, Moscow
  - Novartis Investigational Site, Nizhny Novgorod
  - Novartis Investigational Site, S.-Petersburg
  - Novartis Investigational Site, Saint Petersburg
  - Novartis Investigational Site, Samara
  - Novartis Investigational Site, Smolensk
  - Novartis Investigational Site, Yekaterinburg
- Slovakia (3):
  - Novartis Investigational Site, Banská Bystrica
  - Novartis Investigational Site, Bratislava
  - Novartis Investigational Site, Trnava
- Spain (7):
  - Novartis Investigational Site, Barcelona
  - Novartis Investigational Site, Donostia / San Sebastian
  - Novartis Investigational Site, El Palmar
  - Novartis Investigational Site, Madrid
  - Novartis Investigational Site, Santa Cruz de Tenerife
  - Novartis Investigational Site, Santiago de Compostela
  - Novartis Investigational Site, Valencia
- Sweden (3):
  - Novartis Investigational Site, Gothenburg
  - Novartis Investigational Site, Linköping
  - Novartis Investigational Site, Umeå
- Switzerland (7):
  - Novartis Investigational Site, Aarau
  - Novartis Investigational Site, Carouge
  - Novartis Investigational Site, Geneva
  - Novartis Investigational Site, Lausanne
  - Novartis Investigational Site, Lugano
  - Novartis Investigational Site, Sankt Gallen
  - Novartis Investigational Site, Zurich
- Turkey (Türkiye) (5):
  - Novartis Investigational Site, Antalya
  - Novartis Investigational Site, Gaziantep
  - Novartis Investigational Site, Istanbul
  - Novartis Investigational Site, Samsun
  - Novartis Investigational Site, Trabzon
- United Kingdom (19):
  - Novartis Investigational Site, Birmingham
  - Novartis Investigational Site, Brighton
  - Novartis Investigational Site, Dundee
  - Novartis Investigational Site, Edinburgh
  - Novartis Investigational Site, Essex
  - Novartis Investigational Site, Great Yarmouth
  - Novartis Investigational Site, Headington
  - Novartis Investigational Site, Liverpool
  - Novartis Investigational Site, London
  - Novartis Investigational Site, Middlesbrough
  - Novartis Investigational Site, Newcastle upon Tyne
  - Novartis Investigational Site, Northampton
  - Novartis Investigational Site, Norwick
  - Novartis Investigational Site, Poole
  - Novartis Investigational Site, Salford
  - Novartis Investigational Site, Sheffield
  - Novartis Investigational Site, Stoke-on-Trent
  - Novartis Investigational Site, Swindon
  - Novartis Investigational Site, Truro

REFERENCES:
- [Result] Gold R, Comi G, Palace J, Siever A, Gottschalk R, Bijarnia M, von Rosenstiel P, Tomic D, Kappos L; FIRST Study Investigators. Assessment of cardiac safety during fingolimod treatment initiation in a real-world relapsing multiple sclerosis population: a phase 3b, open-label study. J Neurol. 2014 Feb;261(2):267-76. doi: 10.1007/s00415-013-7115-8. Epub 2013 Nov 13. PMID 24221641